CLINICAL TRIAL: NCT02467127
Title: The Role of Vitamin D Plasma Levels in the Development of Headache
Brief Title: Vitamin D Plasma Level and Its Role in Headache
Acronym: VITDHEAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Catanzaro (Other)
Responsible Party: Principal Investigator, Luca Gallelli, MD, University of Catanzaro
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Headache 2015
Record Dates: First submitted 2015-05-26; First posted 2015-06-09 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Headache
MeSH Terms: conditions — Headache

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- control group (No Intervention): Patients without headache. No drugs will be administered
- Chronic Headache (Experimental): Patients with headache > 6 months. Vitamin D supplementation (from 400 iU/day up to 1600 IU/day) will be administered.
  Interventions: Dietary Supplement: vitamin D supplementation
- Chronic headache with drug overuse (Experimental): Patients with headache > 6 months related to drug treatment, i.e. non steroidal antinflammatory drugs. Vitamin D supplementation (from 400 iU/day up to 1600 IU/day) will be administered.
  Interventions: Dietary Supplement: vitamin D supplementation
- Acute Headache (Experimental): Patients without chronic headache but with an history of headache < 6 months. Vitamin D supplementation (from 400 iU/day up to 1600 IU/day) will be administered.
  Interventions: Dietary Supplement: vitamin D supplementation

INTERVENTIONS:
Dietary Supplement: vitamin D supplementation — In patients with headache and with low vitamin D plasma levels, will be administered a vitamin D supplementation.
  Arms: Acute Headache; Chronic Headache; Chronic headache with drug overuse

SUMMARY:
To date there are conflicting data concerning a correlation between plasma vitamin D levels and headache.

The aim of this study was to evaluate plasma vitamin D levels in patients with headache admitted to the Center of Headache of Pugliese Ciaccio Hospital.

DETAILED DESCRIPTION:
Several papers suggest that inflammation is able to induces both headache and low levels of vitamin D. However, to date a correlation between plasma vitamin D levels and headache has not been demonstrated. Recently we documented that low levels of Vitamin D are related to a low statin efficacy. In this study we will evaluate the plasma levels of vitamin D in patients with headache admitted to the Center of Headache of Pugliese Ciaccio Hospital.

Moreover it will be also evaluated:

* the correlation between efficacy and safety of drugs used in headache treatment and plasma vitamin D levels.
* the role of vitamin D supplementation on both headache symptoms and drug effects.

Plasma vitamin D levels in patients with headache will be evaluated respect to patients without headache.

ELIGIBILITY:
Inclusion Criteria:

* acute or chronic headache diagnosed according to the clinical and radiological criteria of the headache Association

Exclusion Criteria:

* allergy to drugs,
* progressive serious medical conditions (such as cancer, AIDS or end-stage renal disease)
* renal diseases (serum creatinine concentration more than 1.2 times the upper limit of the normal range according to the central laboratory definition reference values)
* liver dysfunction (serum alanine or aspartate transaminase concentrations more than 1.5 times the upper limit of normal range according to the central laboratory definition reference values)
* alcohol consumption (>3 alcoholic beverages daily)
* substance abuse
* inability to give written informed consent
* actual or recent (3-month) treatment with corticosteroids, indomethacin or other antinflammatory drugs.
* secondary headache

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 600 (Actual)
Dates: Start 2015-11; Primary Completion 2017-09 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Plasma levels of vitamin D using high performance liquid chromatography | up to 24 weeks

SECONDARY OUTCOMES:
Headache pain through the Visual Analog Scale (VAS) | up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Luca Gallelli, MD, Principal Investigator — University of Catanzaro
Locations (1):
- Pugliese Hospital, Catanzaro, Italy